CLINICAL TRIAL: NCT01716195
Title: Phase II Trial Of Induction Chemotherapy Followed By Attenuated Chemoradiotherapy For Locally Advanced Head And Neck Squamous Cell Carcinoma Associated With Human Papillomavirus (HPV)
Brief Title: Induction Chemotherapy Followed by Chemoradiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 359512; CCRO022 (Other: UCD)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Cancer
Keywords: Human Papillomavirus; HPV
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Response Adapted Chemoradiation (Experimental): Paclitaxel 175 mg/m2 + Carboplatin area under curve (AUC) 6 followed by response adapted Radiation Therapy (5 - 6 weeks) + Paclitaxel
  Interventions: Radiation: Induction Chemotherapy followed by Response Adapted Chemoradiation

INTERVENTIONS:
Radiation: Induction Chemotherapy followed by Response Adapted Chemoradiation — All patients receive induction chemotherapy with 2 cycles of paclitaxel and carboplatin followed by response adapted, de-escalated chemoradiation. Patients with a complete or partial response will receive 54 Gy with concurrent paclitaxel and patients with stable disease will receive 60 Gy with concurrent paclitaxel.
  Other Names: Paclitaxel; Carboplatin

SUMMARY:
The purpose of this study is to determine whether human papillomavirus (HPV)-positive head and neck cancer can be treated with a less aggressive regimen of radiation therapy and chemotherapy (paclitaxel) after initially receiving two cycles of chemotherapy (carboplatin/paclitaxel).

DETAILED DESCRIPTION:
Given the toxicity of high dose cisplatin, attention has focused on identifying patients at lower risk for failure who may potentially benefit from less aggressive chemoradiotherapy approaches. HPV-positive Head and Neck Cancer responds favorably to radiation therapy. This has prompted investigators to suggest that patients with these cancers might be "over-treated" and unnecessarily subjected to the toxicity of intensive chemoradiotherapy with excessively high radiation doses.

This study will select patients with HPV-positive Head and Neck cancer for attenuated therapy and may have important implications for individualization of care in the future. The regimen of carboplatin and paclitaxel was selected for the induction chemotherapy phase because of its ease of administration, improved toxicity profile, high rates of dose delivery, and excellent published results showing high response rates and overall survival. This study will use induction chemotherapy primarily as a means to select HPV-positive Head and Neck Cancer patients, who may benefit from significant radiation dose de-intensification in the concurrent chemoradiotherapy phase of treatment. The rationale for this risk-adapted approach to local therapy based on HPV status is to administer effective comprehensive treatment individualized at diagnosis and after assessment of response to induction chemotherapy (for patients with HPV-positive tumors), thus avoiding unnecessary and potentially toxic treatment, and hence optimizing the therapeutic ratio.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of HPV-positive squamous cell carcinoma of the oropharynx, hypopharynx, or larynx. HPV-positivity will be defined as tumors that are p16-positive by immunohistochemistry.
* Clinical stage III or IV disease; Note: Patients with M1 tumors are not eligible.
* Appropriate stage for protocol entry, including no distant metastases, based upon minimum diagnostic workup
* Zubrod Performance Status 0-1
* Age > 18
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* Pregnancy test within 4 weeks prior to registration for women of childbearing potential
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study (until at least 60 days following the last study treatment)
* Patient must sign study specific informed consent prior to study entry.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years;
* Patients with simultaneous primaries or bilateral tumors are excluded.
* Patients who present with a cervical lymph node metastasis of unknown primary origin;
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
* Prior radiotherapy that would result in overlap of radiation therapy fields;
* Primary site of tumor of oral cavity, nasopharynx, nasal cavity, paranasal sinuses, or salivary glands;
* Recurrent head and neck cancer;
* Severe, active co-morbidity
* Pregnant or lactating women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Prior allergic reaction to the study drug(s) involved in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2017-03-08 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Daly, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- [Derived] Chen AM, Felix C, Wang PC, Hsu S, Basehart V, Garst J, Beron P, Wong D, Rosove MH, Rao S, Melanson H, Kim E, Palmer D, Qi L, Kelly K, Steinberg ML, Kupelian PA, Daly ME. Reduced-dose radiotherapy for human papillomavirus-associated squamous-cell carcinoma of the oropharynx: a single-arm, phase 2 study. Lancet Oncol. 2017 Jun;18(6):803-811. doi: 10.1016/S1470-2045(17)30246-2. Epub 2017 Apr 20. PMID 28434660

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Response Adapted Chemoradiation
Started | 18
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Response Adapted Chemoradiation
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 63.1 [40.5 to 73.1]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject withdrew consent during treatment phase
  Participants
    number analyzed (Participants) | 17
    Female | 0
    Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject withdrew consent during treatment phase
  Participants
    number analyzed (Participants) | 17
    Hispanic or Latino | 1
    Not Hispanic or Latino | 16
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject withdrew consent during treatment
  Participants
    number analyzed (Participants) | 17
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 17
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival
Description: Defined from date of registration to date of first documentation of progression and/or distant metastasis, or death due to any cause. The true 2-year progression-free survival rate will be estimated by the proportion of efficacy-evaluable patients on study without documentation of disease progression or death 2 years from registration. A 95% confidence interval (CI) for the true progression-free survival rate will be constructed using the Duffy-Santner approach. However, Kaplan-Meier methodology will be used to estimate the final 2-year progression-free survival rate and its 95% CI in case there are censored patients.
Time Frame: Up to 2 years
Population: One subject withdrew consent prior to completing study
Measure: Count of Participants; unit: Participants
Arm/Group | Response Adapted Chemoradiation
Number analyzed (Participants) | 17
Participants | 17

2. Secondary Outcome: Number of Participants With Overall Survival
Description: Defined as the time from registration to death using the Kaplan-Meier method..
Time Frame: Up to 5 years
Population: One subject withdrew consent prior to completing study.
Measure: Count of Participants; unit: Participants
Arm/Group | Response Adapted Chemoradiation
Number analyzed (Participants) | 17
Participants | 16

3. Secondary Outcome: Number of Patients With Toxicity of Concurrent Chemoradiotherapy
Description: Assessed by NCI Common Toxicity Criteria for Adverse Effects, Version 4.0. Reported participants who experienced an AE during concurrent chemoradiotherapy.
Time Frame: Up to 5 years
Population: One subject withdrew consent prior to completing study.
Measure: Count of Participants; unit: Participants
Arm/Group | Response Adapted Chemoradiation
Number analyzed (Participants) | 17
Participants | 17

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Response Adapted Chemoradiation
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Response Adapted Chemoradiation (N=18)
Skin Infection (Infections and infestations) | 1 (1) — MRSA cellulitis
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Dysphagia (General disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Response Adapted Chemoradiation (N=18)
Fatigue (General disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 13
Lymphocyte count decreased (Blood and lymphatic system disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2
Alanine aminotransferase increased (Hepatobiliary disorders) | 3
Aspartate aminotransferase increased (Hepatobiliary disorders) | 3
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 8
White blood cell decreased (Blood and lymphatic system disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Tinnitus (Ear and labyrinth disorders) | 3
Dysphagia (Gastrointestinal disorders) | 8
Dysgeusia (Gastrointestinal disorders) | 5
Sore throat (Gastrointestinal disorders) | 5
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 7
Diarrhea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Oral Pain (Gastrointestinal disorders) | 5
Alkaline phosphatese increased (Hepatobiliary disorders) | 2
Neutrophil count decreased (Immune system disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Myalgia (General disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 4
Sinus bradycardia (Cardiac disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Gastroesophageal reflux disorder (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-02-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT01716195/Prot_SAP_ICF_000.pdf